CLINICAL TRIAL: NCT00080522
Title: Safeguard the Household: A Study of HIV Antiretroviral Therapy Treatment Strategies Appropriate for a Resource Poor Country
Brief Title: Strategies for Delivering Anti-HIV Therapy in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 5U19AI053217-02 (NIH); CIPRA-SA Project 1; 5U19AI053217-02 (NIH)
Record Dates: First submitted 2004-04-06; First posted 2004-04-07 (Estimated); Last update posted 2007-09-18 (Estimated); Status verified 2007-08

CONDITIONS: HIV Infections
Keywords: Treatment Naive; Resource Poor Setting; Drug Delivery; Household; South Africa
MeSH Terms: conditions — HIV Infections | interventions — Stavudine; Lamivudine; efavirenz; Zidovudine; Didanosine; Lopinavir

INTERVENTIONS:
Behavioral: Monitoring by HIV-trained primary care nurses
Behavioral: Community-based directly observed therapy (DOT)
Drug: stavudine
Drug: lamivudine
Drug: efavirenz
Drug: zidovudine
Drug: didanosine
Drug: lopinavir/ritonavir

SUMMARY:
Providing effective anti-HIV therapy in developing countries is challenging. This study will evaluate new strategies for delivering anti-HIV medications to people in South Africa. These strategies include using specially trained nurses to administer therapy (rather than doctors), treating all HIV infected members of a household at the same time, and having community members observe patients taking their medications.

DETAILED DESCRIPTION:
The benefit of antiretroviral therapy is well established but limited to wealthy nations. A predefined, simple sequence of treatment regimens focused on extending the durability of limited treatment options has the best potential to be implemented in resource poor countries. South Africa has 15% of the world's HIV/AIDS patients and a limited number of physicians to treat them (l per 1,600 and less than 5 infectious diseases specialists). HIV patient care in the primary care setting must therefore be delivered by personnel other than doctors. Further, treatment strategies should include entire households to ensure maximum adherence and minimize sharing of drugs.

This study will have two parts. The first part will compare a first-line antiretroviral therapy regimen administered and monitored by primary health care sisters (nurses) with the same regimen administered by doctors. The second part of the study will determine if community-based directly observed therapy (DOT) is significantly superior to continued clinic-based treatment support for patients who have failed first-line therapy, as measured by cumulative virology failure rate. The project will also evaluate the cost and economic impact of a predetermined schedule of antiretroviral therapy; treatment outcomes in terms of morbidity, opportunistic and endemic infections, and mortality; and factors contributing to treatment failure, including toxicity, resistance, compliance, and treatment interruption.

In Part 1, households will be randomly assigned to receive first-line antiretroviral therapy under the monitoring and care of either an HIV-trained medical doctor supported by adherence counselors or an HIV-trained primary health care sister (nurse with training in diagnosis and treatment prescription). Members of the household who are HIV infected will receive stavudine, lamivudine, and efavirenz (nevirapine or nelfinavir may be used for special populations).

Participants who fail first-line antiretroviral therapy in Part 1 of the study will be entered into Part 2 of the study. Participants in Part 2 will receive zidovudine, didanosine, and lopinavir/ritonavir. Participants will be randomly assigned to have their treatment monitored through either a clinic-based treatment support group or through community-based directly observed treatment (DOT). For the DOT arm, a community member will observe therapy for at least one dose a day, five days a week, at the home or work of the participant.

HIV infected children age 3 months to 16 years who live in a participating household will also be included in the study. These children will receive first-line treatment with clinic visits monitored by either the assigned sister (nurse) or doctor along with their households. In Part 2, children will be provided with a second-line treatment regimen with continued daily monitoring of doses in the household.

The study will last 5 years.

ELIGIBILITY:
Inclusion Criteria for the first person in the household who enters the study:

* HIV infected
* Older than 16 years of age
* History of a severe CDC Category B or C AIDS-defining illness or a CD4 cell count less than 350 cells/mm3 within 6 months prior to study entry
* Have not previously taken anti-HIV medications. People who have taken anti-HIV medications for post-exposure prophylaxis or prevention of mother-to-child transmission may be eligible if the previous exposure did not exceed 6 weeks of nucleoside reverse transcriptase inhibitors or protease inhibitors, or two doses of a non-nucleoside reverse transcriptase inhibitor.

Inclusion Criteria for children between 3 and 16 years old in a household that has been entered in the study:

* HIV infected
* Live in house with an adult participating in the study
* History of severe CDC Category B or C AIDS-defining illness, with the exception of a single episode of bacterial sepsis or a single episode of Zoster; or one CD4% less than 20% (less than 25% for children 3 to 18 months) obtained within 6 months prior to study entry
* Have not previously taken anti-HIV medications. Children who have taken anti-HIV medications for post-exposure prophylaxis or prevention of mother-to-child transmission may be eligible if the previous exposure did not exceed 6 weeks of nucleoside reverse transcriptase inhibitors or protease inhibitors, or two doses of a non-nucleoside reverse transcriptase inhibitor therapy. Children who received 6 weeks of AZT or a single dose of nevirapine will be included in the study.
* Consent of parent or legal guardian
* Primary caregiver who is willing and able to administer anti-HIV medications

Exclusion Criteria:

* Newly diagnosed AIDS-defining (CDC Classification C) opportunistic infection or condition requiring acute therapy at the time of enrollment. A stable patient on therapy for more than 7 days may be enrolled. Patients who tuberculosis treatment within 8 weeks of the baseline visit are not excluded.
* Use of medications with significant effect on bone marrow, nervous system, pancreas, or liver within 30 days prior to study entry
* Use of cytotoxic medications within 30 days prior to study entry
* Active alcohol or substance abuse
* Severe diarrhea (more than 6 stools/day for 7 consecutive days) within 30 days prior to study entry
* Acute hepatitis within 30 days prior to study entry
* Bilateral peripheral neuropathy of Grade 2 or greater at the time of screening
* Women in the first trimester of pregnancy
* Women who have failed a lopinavir/ritonavir treatment regimen in Part I and who are either pregnant at entry into Part 2 or are of childbearing potential with a CD4 count of 250 cells/mm3 or more
* Inability to tolerate oral medication
* Any clinical condition that, in the opinion of the investigator, would make the person unsuitable for the study or unable to comply with the dosing requirements

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 813
Dates: Start 2005-02; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Cumulative treatment failure rate, determined by comparing a primary health care level first line antiretroviral therapy regimen to a doctor monitored treatment regimen
48-week cumulative virology failure rate, determined by comparing community-based directly observed therapy (DOT) by identified and trained community members to continued clinic-based treatment support for subjects who have failed first line therapy

SECONDARY OUTCOMES:
Overall clinical safety of antiretroviral therapy, as measured by the occurrence of clinical and laboratory Grade 3 and 4 adverse events, between primary health care monitoring arms in adults and children
CD4+ count, viral load, drug toxicity, adherence, participation in MTCT programs, intercurrent medical conditions, age as factors potentially contributing to cumulative treatment failure in participants age 16 and older
cumulative treatment failure rate between groups, defined by clinical staging (CDC and WHO classification) prior to initiation of antiretroviral therapy and monitoring arms in adults and children
cumulative treatment failure rate of second line therapy from time of Phase 1 randomization in adults and children, between the doctor and the primary health care sister-based monitoring arm
comparison of immune reconstitution in adults and children, using change in CD4+ percent from baseline between the two treatment monitoring models over the duration of the study
comparison of HIV resistance mutations in adults and children who have demonstrated virologic failure between the doctor and the primary health care sister-based monitoring arms
comparison of adherence to antiretroviral treatment in Phase 1 in both adults and children as measured by pill count (or weight or volume of drug solution) between the two primary health care monitoring models
comparison of adherence to antiretroviral treatment in adults as measured by pill count between those randomized to community-based DOT and those randomized to continued clinic-based adherence support
comparison of HIV disease progression/death in adults and children between the two primary health care monitoring arms
total and incremental costs of adding the 4 approaches for the provision of antiretrovirals to primary health care services in each study site
potential costs to the government of provincial and national based scale-up for the provision of antiretroviral therapy in the short, long and medium term and resulting net costs/savings of each approach as a national strategy
relative cost effectiveness of the introduction of the four alternative models of HAART provision versus no provision, using life-years gained and quality adjusted life-years gained
household preferences for various aspects of antiretroviral therapy provision program design, including assessing their relationship with adherence
personnel required for a nurse-based monitoring program, including the training process and implementation

CONTACTS AND LOCATIONS:
Locations (2):
- South Africa (2):
  - University of the Witwatersrand/Clinical HIV Research Unit, Johannesburg, Gauteng
  - University of Cape Town/Masiphumelele, Cape Town, South Peninsula